CLINICAL TRIAL: NCT07341958
Title: INtensive liPid-lowering Therapy for Acute High-risk IntracRanial or Extracranial atheroSclerosis -II (INSPIRES-2)：A Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: INtensive liPid-lowering Therapy for Acute High-risk IntracRanial or Extracranial atheroSclerosis -II (INSPIRES-2)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, yilong Wang, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HX-A-2025103
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Ischemic Stroke or High-risk TIA (ABCD² ≥ 4)
Keywords: PCSK9 inhibitor; lipid-lowering therapy; ischemic stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: A multicenter, randomized, double-blind, placebo-controlled clinical trial
Who Masked: Participant, Investigator
Masking Description: The active drug and placebo are identical in appearance, packaging, labeling, and administration. Standard background lipid-lowering therapy (statin ± ezetimibe) is administered to both groups and does not affect blinding. Routine tests and imaging at study sites contain no group allocation information, preventing unintentional unblinding. Investigators and subjects must remain blinded to treatment assignment. Unblinding of randomization codes is prohibited unless required for managing a serious adverse event (SAE). All unblinding events must be fully documented and reported to the sponsor and the independent Data Safety Monitoring Board (DSMB).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard lipid-lowering therapy(statin therapy with or without ezetimibe) + Tafolecimab (Experimental)
  Interventions: Drug: Tafolecimab
- Standard lipid-lowering therapy (statin therapy with or without ezetimibe)+Tafolecimab placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tafolecimab — Treatment should be initiated as soon as possible after randomization, with Tafolecimab administered subcutaneously once every two weeks for a total duration of 90 days.
  All patients received standard lipid-lowering therapy as recommended by stroke secondary prevention guidelines, including intensive statin treatment with or without ezetimibe, administered at maximally tolerated doses.
  Arms: Standard lipid-lowering therapy(statin therapy with or without ezetimibe) + Tafolecimab
Drug: Placebo — Treatment should be initiated as soon as possible after randomization, with Tafolecimab placebo administered subcutaneously once every two weeks for a total duration of 90 days.
  All patients received standard lipid-lowering therapy as recommended by stroke secondary prevention guidelines, including intensive statin treatment with or without ezetimibe, administered at maximally tolerated doses.
  Arms: Standard lipid-lowering therapy (statin therapy with or without ezetimibe)+Tafolecimab placebo

SUMMARY:
The research team is conducting a randomized, double-blind, placebo-controlled, multicenter clinical study aimed at evaluating the impact of adding Tolecilimab (a PCSK9 inhibitor) to standard lipid-lowering therapy (statins ± ezetimibe) on serum lipoprotein(a) [Lp(a)] levels and the risk of stroke recurrence within 90 days in patients with ischemic stroke or high-risk TIA (ABCD² ≥ 4) accompanied by elevated lipoprotein(a) levels (≥50 mg/dL).

DETAILED DESCRIPTION:
Atherosclerotic stroke, particularly the large-artery atherosclerosis (LAA) subtype, carries a high risk of recurrence despite standard lipid-lowering therapy with statins. Elevated Lipoprotein(a) [Lp(a)] is a key genetic, pro-atherogenic risk factor largely unaffected by conventional statins and is independently associated with an increased risk of LAA-type stroke recurrence, representing a significant unmet residual risk. Proprotein convertase subtilisin/kexin type 9 (PCSK9) inhibitors provide a dual-pathway approach by potently lowering both low-density lipoprotein cholesterol (LDL-C) and Lp(a) levels.Evidence on the benefits of early, intensive lipid-lowering with PCSK9 inhibitors specifically for secondary stroke prevention in high-risk LAA patients with elevated Lp(a) is lacking. The primary purpose of this study is to evaluate the efficacy and safety of adding tafolecimab, a novel PCSK9 inhibitor, to standard lipid-lowering therapy in reducing Lp(a) levels at 90 days in patients with acute ischemic stroke or high-risk transient ischemic attack (TIA) of LAA etiology and elevated Lp(a). Secondary objectives include assessing its impact on LDL-C control, preliminary clinical outcomes (stroke recurrence, composite vascular events), safety, and exploring biomarker associations. This is a multicenter, randomized, double-blind, placebo-controlled clinical trial. A total of 242 patients from multiple centers in China will be enrolled. Key eligibility criteria include: age 35-80 years, acute ischemic stroke or high-risk TIA (ABCD² ≥4) of large-artery atherosclerosis (LAA) etiology occurring 3-7 days before randomization, and lipoprotein(a) [Lp(a)] ≥50 mg/dL. Patients will be stratified by site and randomly assigned in a 1:1 ratio to receive either standard lipid-lowering therapy (statin ± ezetimibe) plus tafolecimab (a PCSK9 monoclonal antibody) or standard therapy plus matching placebo for 90 days. Study treatment will be initiated as soon as possible after randomization. Face-to-face visits are scheduled at baseline, day 7 (or hospital discharge), and months 1, 2, and 3 after randomization. At each visit, neurological status (NIHSS, mRS), vital signs, concomitant medications, and adverse events will be recorded. Fasting blood samples will be collected at baseline, month 1, month 2, and month 3 for central laboratory measurement of Lp(a), LDL-C, apolipoprotein B, high-sensitivity C-reactive protein, and interleukin-6. Additional safety laboratories (liver function, renal function, creatine kinase, complete blood count) will be performed at baseline, day 7, and month 3. The primary efficacy endpoint is the percent change in Lp(a) from baseline to 90 days, analyzed using a repeated-measures mixed-effects model (MMRM) with adjustment for baseline value. The key secondary efficacy endpoints include: percent change in LDL-C at 90 days, proportion of patients achieving LDL-C goal (<1.8 mmol/L or ≥50% reduction), and the occurrence of stroke recurrence, composite vascular events (ischemic stroke, myocardial infarction, hospitalization for unstable angina or heart failure, cardiovascular death), and all-cause death within 90 days. Safety endpoints comprise the incidence of adverse events, serious adverse events, bleeding events (GUSTO classification), hepatotoxicity (ALT/AST >3× ULN), myotoxicity (CK >10× ULN or clinical muscle symptoms), and injection-site reactions. The sample size was calculated to provide 80% power to detect a 25% between-group difference in Lp(a) reduction at 90 days, assuming a standard deviation of 67.34% and a two-sided alpha of 0.05, with an anticipated 5% dropout rate. Efficacy analyses will be performed on the intention-to-treat (ITT) population, while safety analyses will include all patients who received at least one dose of study drug. Time-to-event endpoints will be analyzed using Kaplan-Meier estimates and Cox proportional-hazards models. Continuous secondary endpoints will be assessed using MMRM or analysis of covariance.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 35 and 80 years, regardless of gender.
2. For patients with prior lipid-lowering treatment: screening LDL-C ≥1.8 mmol/L; for treatment-naïve patients: screening LDL-C ≥2.6 mmol/L.
3. Lp(a) ≥50 mg/dL.
4. Onset of symptoms within 3 to 7 days.
5. Diagnosis of ischemic stroke (NIHSS score ≤20) or high-risk TIA with ABCD² score ≥4; and meeting at least one of the following imaging criteria:

(1) Large-artery atherosclerosis (LAA) subtype per TOAST classification: vascular imaging confirms ≥50% atherosclerotic stenosis of the intracranial or extracranial culprit artery.

(2) Head CT or MRI demonstrates acute multiple infarcts, with etiology consistent with large-artery atherosclerosis (including nonstenotic vulnerable plaques).

6.The patient or their legally authorized representative has provided written informed consent.

Exclusion Criteria:

1. Patients who have undergone or are scheduled to undergo thrombolysis or thrombectomy therapy.
2. Definite cardiogenic ischemic cerebrovascular disease (e.g., accompanied by atrial fibrillation, prosthetic heart valves, atrial myxoma, infective endocarditis, etc.).
3. Other clearly identified etiologies of ischemic cerebrovascular disease (e.g., aortic dissection, cervical/cerebral arterial dissection, vasculitis, vascular malformations, moyamoya disease/syndrome, fibromuscular dysplasia, etc.).
4. Non-vascular intracranial diseases (e.g., intracranial tumors, multiple sclerosis, etc.).
5. Imaging findings indicating that the current cerebral infarction area exceeds 1/2 of a single brain lobe.
6. Imaging findings indicating hemorrhagic transformation of the current cerebral infarction.
7. Pre-stroke mRS score > 2.
8. Patients with known allergies to Tafolecimab or other contraindications for its use.
9. Use of immunosuppressive drugs, antifungal drugs, or fibrates (which affect statin metabolism) within 14 days prior to randomization.
10. Creatine kinase levels exceeding 5 times the upper limit of normal after the onset of the event.
11. Severe hepatic or renal insufficiency prior to randomization (Note: Severe hepatic insufficiency is defined as ALT >2×ULN or AST >2×ULN; severe renal insufficiency is defined as serum creatinine >1.5×ULN or GFR <40 ml/min/1.73m²).
12. History of intracranial hemorrhage (e.g., ICH, SAH).
13. History of intracranial or extracranial vascular angioplasty.
14. History of gastrointestinal bleeding or major surgery within 90 days prior to enrollment.
15. Planned surgical or interventional procedures within the next 90 days that may necessitate discontinuation of the investigational drug.
16. Suffering from severe organic diseases with an expected survival time of less than 1 year.
17. Pregnant women, or women of childbearing potential who are not using effective contraception and lack documented pregnancy test results.
18. Currently participating in other investigational drug or device trials.
19. Inability to cooperate with follow-up due to geographic, social, or other reasons (e.g., alcohol abuse, substance abuse, dementia, severe psychiatric disorders, etc.).

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
The percentage reduction in Lp(a) from baseline at 90 days. | From baseline to 90 days after randomization

SECONDARY OUTCOMES:
Incidence of new stroke (including hemorrhagic and ischemic stroke) within 90 days. | From baseline to 90 days after randomization
  Symptoms and signs of acute neurological deficits caused by sudden focal or whole brain, spinal cord or retinal vascular damage, which are related to cerebral circulatory disorders, including hemorrhagic and ischemic stroke
Incidence of composite clinical endpoint events within 90 days | From baseline to 90 days after randomization
  Including recurrent ischemic stroke, myocardial infarction, rehospitalization for unstable angina or heart failure, and cardiovascular death
Incidence of myocardial infarction within 90 days. | From baseline to 90 days after randomization
  Acute myocardial infarction is diagnosed by the third edition of the international general diagnostic criteria (Glob Heart. 2012 Dec;7(4):275-95)
Incidence of vascular death within 90 days. | From baseline to 90 days after randomization
  Vascular death includes stroke, sudden cardiac death, acute myocardial infarction, heart failure, pulmonary embolism, heart / cerebrovascular intervention or surgery (death unrelated to acute MI) and other cardiovascular causes of death [such as: Arrhythmia irrelevant with sudden cardiac death, aortic aneurysm rupture, or peripheral artery disease. Any death of unknown/unclear cause that occurs within 30 days after stroke, myocardial infarction, or cardio-cerebrovascular operation/surgery will be regarded as death due to stroke, myocardial infarction, or cardio-cerebrovascular operation/surgery, respectively.
Incidence of all-cause death within 90 days. | From baseline to 90 days after randomization
Proportion of patients with poor functional outcome (mRS score 2-6) at 90 days. | From baseline to 90 days after randomization
  The Modified Rankin Scale (mRS) score ranges from 0 to 6, with higher scores indicating worse functional outcome. The modified Rankin Scale (mRS)= 2-6: poor functional outcome
Proportion of patients with Lp(a) <30 mg/dL at 90 days | From baseline to 90 days after randomization
Percent reduction in ApoB and LDL-C levels from baseline to 90 days | From baseline to 90 days after randomization
LDL-C goal attainment rate (<1.8 mmol/L or reduction ≥ 50%) at 90 days | From baseline to 90 days after randomization
Moderate and severe bleeding events (GUSTO classification) | From baseline to 90 days after randomization
  The GUSTO classification provides a three-tiered (severe, moderate, mild), criteria-driven framework for consistently reporting bleeding complications in clinical research, with a focus on hemodynamic impact and objective laboratory/transfusion data.
Hepatotoxicity: Post-treatment ALT or AST levels exceeding 3 times the upper limit of normal upon re-measurement | From baseline to 90 days after randomization
  Hepatotoxicity in this context is defined as a confirmed elevation of liver enzymes after treatment. Specifically, it means that a follow-up blood test shows either ALT or AST levels to be more than three times higher than the normal limit. This is a standard safety criterion for detecting potential drug-induced liver injury in clinical trials.
Muscle toxicity | From baseline to 90 days after randomization
  Post-treatment creatine kinase levels exceeding 10 times the upper limit of normal upon re-measurement, or occurrence of skeletal muscle adverse events (myalgia, myopathy, or rhabdomyolysis)
Upper Respiratory Tract Infection (URTI): | From baseline to 90 days after randomization
  Common infections affecting the nose, sinuses, throat, or larynx (e.g., common cold, sinusitis). These are general illnesses, not necessarily treatment-related.
Urinary Tract Infection (UTI) | From baseline to 90 days after randomization
  An infection in any part of the urinary system (bladder, urethra, kidneys). It is monitored as a common potential infection during trials.
Injection Site Reactions: | From baseline to 90 days after randomization
  Including papules, bleeding, discoloration, pain, itching, rash, induration, erythema, swelling, etc., at the injection site
Allergic Reactions: | From baseline to 90 days after randomization
  Undesirable immune system responses to the treatment, ranging from mild (rash, itching) to severe, life-threatening anaphylaxis.
Other Adverse Events/Serious Adverse Events (AEs/SAEs): | From baseline to 90 days after randomization
  Other Adverse Events/Serious Adverse Events (AEs/SAEs):

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hopital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No